CLINICAL TRIAL: NCT05048433
Title: Developing and Testing an Implementation Strategy for Active Learning to Promote Physical Activity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Timothy J Walker, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-20-0861; K01HL151817 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Physical Activity
Keywords: Implementation of Physical Activity Programs in Schools
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation strategy for active learning to promote physical activity (Experimental)
  Interventions: Behavioral: Implementation strategy for active learning to promote physical activity
- Usual implementation support (Active Comparator)
  Interventions: Behavioral: Usual implementation support

INTERVENTIONS:
Behavioral: Implementation strategy for active learning to promote physical activity — The experimental arm includes using a multifaceted implementation strategy to support the use of classroom-based physical activity approaches. The strategy consists of a series of leadership trainings designed to help them support teachers, teacher trainings to build skills, and a monthly newsletter to reinforce implementation and provide access to existing resources.
  Arms: Implementation strategy for active learning to promote physical activity
Behavioral: Usual implementation support — Usual support consists of the potential to access general resources from the district wellness department. These resources include access to funds to send staff to external trainings and general guidance for how to use active learning approaches.
  Arms: Usual implementation support

SUMMARY:
The purpose of this study is to develop an implementation strategy to improve the use and sustainment of active learning in elementary schools and to conduct a feasibility study to evaluate the impact of the developed implementation strategy on the implementation and effectiveness of active learning.

ELIGIBILITY:
Inclusion Criteria:

* lead teachers who teach kindergarten to fifth grade
* children in kindergarten to fifth grade

Exclusion Criteria:

* non English or Spanish speaking

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Walker, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walker TJ, Craig DW, Pfledderer CD, Lee M, Onadeko K, Saving EE, Bartholomew JB, Fernandez ME. Feasibility and acceptability of an implementation strategy to enhance use of classroom-based physical activity approaches in elementary schools: a mixed methods study. BMC Public Health. 2025 Nov 27;26(1):36. doi: 10.1186/s12889-025-25333-0. PMID 41310531
- [Derived] Walker TJ, Kohl HW 3rd, Bartholomew JB, Green C, Fernandez ME. Using Implementation Mapping to develop and test an implementation strategy for active learning to promote physical activity in children: a feasibility study using a hybrid type 2 design. Implement Sci Commun. 2022 Mar 7;3(1):26. doi: 10.1186/s43058-022-00271-9. PMID 35256018

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: School
Period: Fall 2023
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Started | 136; 1 School | 133; 1 School
Children | 106; 1 School | 101; 1 School
Teachers | 30; 1 School | 32; 1 School
Completed | 136; 1 School | 133; 1 School
Not Completed | 0; 0 School | 0; 0 School
Period: Spring 2024
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Started | 136; 1 School | 134; 1 School (1 New teacher enrolled in the Usual Implementation support arm during the Spring 2024 period.)
Children | 106; 1 School | 101; 1 School
Teachers | 30; 1 School | 33; 1 School (1 New teacher enrolled in the Usual Implementation support arm during the Spring 2024 period.)
Completed | 136; 1 School | 134; 1 School
Not Completed | 0; 0 School | 0; 0 School
Period: Fall 2024
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Started | 129; 1 School | 118; 1 School
Children | 104; 1 School (Of the 106 children enrolled in Fall 2023 in the Implementation strategy for active learning to promote physical activity arm , 18 new students were added and 20 students left, resulting in 104 children enrolled in Fall 2024) | 92; 1 School (Of the 101 children enrolled in Fall 2023 in the Usual implementation support arm arm , 3 new students were added and 12 students left, resulting in 92 children enrolled in Fall 2024)
Teachers | 25; 1 School (Of the 30 teachers enrolled in Fall 2023 in the Implementation strategy for active learning to promote physical activity arm, 5 new teachers were added and 10 teachers left, resulting in 30 teachers enrolled in Fall 2024) | 26; 1 School (Of the 33 teachers enrolled in Spring 2024 in the Usual implementation support arm, 5 new teachers were added and 12 teachers left, resulting in 26 teachers enrolled in Fall 2024.)
Completed | 129; 1 School | 118; 1 School
Not Completed | 0; 0 School | 0; 0 School

BASELINE CHARACTERISTICS:
Population: 159 participants (124 children and 35 teachers) were assigned to the Implementation strategy for active learning to promote physical activity arm. 142 participants (38 teachers and 104 children) were assigned to the Usual implementation support arm. The number shown in each group reflect unique participants (both teachers and children).
Groups:
- Total: Total of all reporting groups
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support | Total
Number analyzed (Participants) | 159 | 142 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data were not collected from 6 Teacher participants in the Usual implementation support arm because 3 teacher participants did not complete the survey and 3 did not answer this question. Baseline data were not collected for 1 child participant in each arm because the study team was unable to obtain the required information from the school partners. As a result, these participants were not included in the baseline analysis for age.
  years
    Children: number analyzed (Participants) | 123 | 103 | 226
    Children | 7.6 (1.4) | 7.3 (1.5) | 7.5 (1.5)
    Teachers: number analyzed (Participants) | 35 | 32 | 67
    Teachers | 35.4 (11) | 41.9 (12.6) | 38.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were not collected from 6 Teacher participants in the Usual implementation support arm because 3 teacher participants did not complete the survey and 3 did not answer this question. Baseline data were not collected for 1 child participant in each arm because the study team was unable to obtain the required information from the school partners. As a result, these participants were not included in the baseline analysis for sex: Female, Male.
  Participants
    Children: number analyzed (Participants) | 123 | 103 | 226
    Children: Female | 57 | 54 | 111
    Children: Male | 66 | 49 | 115
    Teachers: number analyzed (Participants) | 35 | 32 | 67
    Teachers: Female | 31 | 23 | 54
    Teachers: Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 159 participants (124 children and 35 teachers) were assigned to the Implementation strategy for active learning to promote physical activity arm. 142 participants (38 teachers and 104 children) were assigned to the Usual implementation support arm. The number shown in each group reflect unique participants (both teachers and children).
  Participants
    Children: number analyzed (Participants) | 124 | 104 | 228
    Children: Hispanic or Latino | 71 | 72 | 143
    Children: Not Hispanic or Latino | 52 | 31 | 83
    Children: Unknown or Not Reported | 1 | 1 | 2
    Teachers: number analyzed (Participants) | 35 | 38 | 73
    Teachers: Hispanic or Latino | 8 | 14 | 22
    Teachers: Not Hispanic or Latino | 27 | 18 | 45
    Teachers: Unknown or Not Reported | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 159 participants (124 children and 35 teachers) were assigned to the Implementation strategy for active learning to promote physical activity arm. 142 participants (38 teachers and 104 children) were assigned to the Usual implementation support arm. The number shown in each group reflect unique participants (both teachers and children)..
  Participants
    Children: number analyzed (Participants) | 124 | 104 | 228
    Children: American Indian or Alaska Native | 17 | 23 | 40
    Children: Asian | 1 | 3 | 4
    Children: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Children: Black or African American | 41 | 30 | 71
    Children: White | 63 | 46 | 109
    Children: More than one race | 0 | 0 | 0
    Children: Unknown or Not Reported | 1 | 1 | 2
    Teachers: number analyzed (Participants) | 35 | 38 | 73
    Teachers: American Indian or Alaska Native | 1 | 3 | 4
    Teachers: Asian | 0 | 1 | 1
    Teachers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Teachers: Black or African American | 21 | 12 | 33
    Teachers: White | 12 | 12 | 24
    Teachers: More than one race | 1 | 4 | 5
    Teachers: Unknown or Not Reported | 0 | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States | 159 | 142 | 301
Student's Lunch Status [Count of Participants; unit: Participants] — Population: Student's Lunch Status was only measured for the Children (students) participants.
  Participants
    number analyzed (Participants) | 124 | 104 | 228
    Reduced Lunch | 21 | 9 | 30
    Free | 93 | 85 | 178
    Non-participant | 9 | 9 | 18
    Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Active Learning Among Teachers as Assessed by the Acceptability of Implementation Measure (AIM)
Description: The Acceptability of Implementation Measure (AIM) total score is from 1 to 5, with higher scores representing higher levels of acceptability.
Time Frame: Baseline
Population: Data were only collected from Teacher Participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 29 | 27
score on a scale | 4.7 (0.4) | 4.3 (1)

2. Primary Outcome: Acceptability of Active Learning Among Teachers as Assessed by the Acceptability of Implementation Measure (AIM)
Description: as for outcome 1
Time Frame: Approximately 7 months after baseline
Population: Data were only collected from Teacher Participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 30 | 26
score on a scale | 4.6 (0.7) | 4.5 (0.9)

3. Primary Outcome: Acceptability of Active Learning Among Teachers as Assessed by the Acceptability of Implementation Measure (AIM)
Description: as for outcome 1
Time Frame: Approximately 13 months after baseline
Population: Data were only collected from Teacher Participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 24 | 19
score on a scale | 4.7 (0.4) | 4.8 (0.4)

4. Primary Outcome: Implementation Fidelity as Assessed by Self-reported Implementation Logs to Assess Dose of Delivery
Description: Implementation logs will be completed weekly throughout the study and dose of delivery is the number of minutes per day of active learning used.
Time Frame: Baseline
Population: Data were only collected from Teacher Participants who completed the self-reported implementation log.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 21 | 23
minutes per day | 6.5 (8.8) | 6.8 (16.7)

5. Primary Outcome: Implementation Fidelity as Assessed by Self-reported Implementation Logs to Assess Dose of Delivery
Description: Implementation logs will be completed weekly throughout the study and dose of delivery is the number of minutes per week of active learning used.
Time Frame: Approximately 7 months after baseline
Population: Data were only collected from Teacher Participants who completed the self-reported implementation log.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 27 | 24
minutes per day | 13.5 (17.2) | 12.9 (16.8)

6. Primary Outcome: Implementation Fidelity as Assessed by Self-reported Implementation Logs to Assess Dose of Delivery
Description: as for outcome 4
Time Frame: Approximately 13 months after baseline
Population: Data were only collected from Teacher Participants who completed the self-reported implementation log.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 24 | 21
minutes per day | 9.3 (19.5) | 9.7 (9.7)

7. Primary Outcome: Implementation Fidelity as Assessed by Teacher Survey of Dose of Delivery
Description: Dose of delivery is the number of minutes per day of active learning used.
Time Frame: Baseline
Population: Data were only collected from Teacher Participants who completed the Survey.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 29 | 27
minutes per day | 11.8 (10.5) | 8.3 (9.1)

8. Primary Outcome: Implementation Fidelity as Assessed by Teacher Survey of Dose of Delivery
Description: Dose of delivery is the number of minutes per day of active learning used.
Time Frame: Approximately 7 months after baseline
Population: Data were only collected from Teacher Participants who completed the Survey.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 30 | 27
minutes per day | 16 (10.9) | 12.8 (12.6)

9. Primary Outcome: Implementation Fidelity as Assessed by Teacher Survey of Dose of Delivery
Description: Dose of delivery is the number of minutes per day of active learning used.
Time Frame: Approximately 13 months after baseline
Population: Data were only collected from Teacher Participants who completed the Survey.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 24 | 19
minutes per day | 14.5 (11.8) | 14.3 (12.7)

10. Primary Outcome: Student Physical Activity as Indicated by Number of Minutes Per Day Spent in Moderate and Vigorous Physical Activity as Assessed by the Actigraph GT3X+ Accelerometer
Time Frame: Baseline
Population: Data were collected only from participants who wore the ActiGraph GT3X+ accelerometer for sufficient time to meet valid wear-time criteria.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 100 | 97
minutes per day | 26.5 (11.1) | 25.1 (8.9)

11. Primary Outcome: Student Physical Activity as Indicated by Number of Minutes Per Day Spent in Moderate and Vigorous Physical Activity as Assessed by the Actigraph GT3X+ Accelerometer
Time Frame: Approximately 7 months after baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 84 | 82
minutes per day | 25.2 (10.3) | 26.7 (9.8)

12. Primary Outcome: Student Physical Activity as Indicated by Number of Minutes Per Day Spent in Moderate and Vigorous Physical Activity as Assessed by the Actigraph GT3X+ Accelerometer
Time Frame: Approximately 13 months after baseline
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity | Usual Implementation Support
Number analyzed (Participants) | 92 | 88
minutes per day | 22.7 (8.2) | 26.2 (8.7)

ADVERSE EVENTS:
Time Frame: From Fall 2023 to Fall 2024 (About 15 months)
Groups:
- Implementation Strategy for Active Learning to Promote Physical Activity: Children; Implementation Strategy for Active Learning to Promote Physical Activity: Teachers: Implementation strategy for active learning to promote physical activity: The experimental arm includes using a multifaceted implementation strategy to support the use of classroom-based physical activity approaches. The strategy consists of a series of leadership trainings designed to help them support teachers, teacher trainings to build skills, and a monthly newsletter to reinforce implementation and provide access to existing resources.
- Usual Implementation Support: Children; Usual Implementation Support: Teachers: Usual implementation support: Usual support consists of the potential to access general resources from the district wellness department. These resources include access to funds to send staff to external trainings and general guidance for how to use active learning approaches.
Arm/Group | Implementation Strategy for Active Learning to Promote Physical Activity: Children | Usual Implementation Support: Children | Implementation Strategy for Active Learning to Promote Physical Activity: Teachers | Usual Implementation Support: Teachers
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/104 | 0/35 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/104 | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 0/124 | 0/104 | 0/38 | 0/35

LIMITATIONS AND CAVEATS:
The reported implementation and physical activity outcomes are unadjusted values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT05048433/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT05048433/ICF_001.pdf